CLINICAL TRIAL: NCT02193412
Title: Influence of Variations of Systemic Venous Return on Analgesia Nociception Index (ANI) During General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013_13; 2013-A01645-40 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Hypovolemia; Somatic Pain
Keywords: analgesia nociception index; heart rate variability; autonomic nervous system; specificity; systemic venous return; pulse pressure variation; Intraoperative Monitoring
MeSH Terms: conditions — Hypovolemia; Nociceptive Pain | interventions — Head-Down Tilt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients (Experimental): 1. noxious stimulus
  2. change in operating table slope: head-down tilt position
  3. change in operating table slope: head-up tilt position
  Interventions: Procedure: noxious stimulus; Procedure: change in operating table slope: head-down tilt position; Procedure: change in operating table slope: head-up tilt position

INTERVENTIONS:
Procedure: noxious stimulus — standardized noxious stimulus with tetanic stimulation
Procedure: change in operating table slope: head-down tilt position — -30°
  Other Names: Trendelenburg position
Procedure: change in operating table slope: head-up tilt position — +30°

SUMMARY:
The purpose of this study is to determine whether the value of analgesia nociception index (ANI) is influenced by variations of systemic venous return (cardiac preload) under general anaesthesia.

DETAILED DESCRIPTION:
In the context of opioid sparing goal during general anaesthesia, the Analgesia nociception index (ANI) is an analgesia/nociception balance monitoring tool computed from high frequency heart rate variability analysis, and developed by MetroDoloris (Lille, France). Its sensitivity to detect noxious stimulus was studied in several studies. However, its specificity is not established in particular in the presence of factors influencing autonomic nervous system other than analgesia/nociception balance. In the context of anaesthesia, one of the most relevant factor is hypovolemia. This study aims to assess the effect of blood volume variations on ANI under general anaesthesia, independently of analgesia/nociception balance status. Variations of systemic venous return (SVR) (cardiac preload), which reflects blood volume status, will be induced by changes of operating table slope, from head-down tilt (Trendelenburg), with increased SVR, to head-up tilt position, with decreased SVR. Variations of SVR will be attested by changes in the arterial pulse pressure variation, a well-established indice of preload responsiveness in the mechanically ventilated anaesthetized patient.

ELIGIBILITY:
Inclusion Criteria:

* neurosurgical operation requiring invasive monitoring of arterial blood pressure

Exclusion Criteria:

* pacemaker, arrhythmia
* chronic medication with beta blocker
* possible disorder of autonomic nervous system: diabetes, alcoholism, chronic pain
* anticholinergic drug administration before measures
* intracranial hypertension
* no social security coverage
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-04 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
change in ANI between head-down tilt (Trendelenburg) position and head-up tilt position | during changes of operating table slope (i.e., for 1-2 min in each condition, 10-15 min after initial measurements in basal conditions)
  Position -20° to +20°

SECONDARY OUTCOMES:
change in ANI between horizontal position and head-down/head up tilt position | during changes of operating table slope (i.e., for 1-2 min in each condition, 10-15 min after initial measurements in basal conditions)
  Position 0° to -20° Position +20° to 0°
change in pulse pressure variation between head-down tilt position and head-up tilt position | during changes of operating table slope (i.e., for 1-2 min in each condition, 10-15 min after initial measurements in basal conditions)
  Position -20° to +20°
change in ANI induced by standardized noxious stimulus (tetanic stimulation) | during a 5sec-tetanic stimulation (measurement for 1-2 min, 2-5 min after initial measurements in basal conditions)
  ANI measurement following tetanus
variations of low frequency variability of arterial blood pressure | during changes of operating table slope (i.e., for 1-2 min in each condition, 10-15 min after initial measurements in basal conditions)
  Position 0° to -20° Position -20° to +20° Position +20° to 0°
change in pulse pressure variation between horizontal position and head-down/head up tilt position | during changes of operating table slope (i.e., for 1-2 min in each condition, 10-15 min after initial measurements in basal conditions)
  Position 0° to -20° Position +20° to 0°

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Tavernier, Pr, Principal Investigator — Lille University Hospital; Délégation à la Recherche Clinique et à l'Innovation (DRC), Study Chair — Lille University Hospital
Locations (1):
- University Hospital, Lille, Nord, France